CLINICAL TRIAL: NCT05937217
Title: Quality of Life and Pain Pressure Threshold in Response to Myofascial Induction Therapy and Direct Scar Release Techniques for Chronic Lower Transverse Abdominal Scar
Brief Title: Quality of Life and Pain Pressure Threshold in Response to Scar Release Techniques for Chronic Transverse Abdominal Scar
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, manal ahmed el-shafei mohamed, lecturer of physical therapy for women's health , faculty of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004580
Record Dates: First submitted 2023-06-30; First posted 2023-07-10 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Cesarean Section Complications
MeSH Terms: interventions — Ultrasonic Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- myofascial induction and direct scar release techniques group (Experimental): They will receive myofascial induction therapy in the form of transverse sliding and cross hand therapy and direct scar release techniques in the form of stroking, circular movement, vertical point lifting , C and S grip techniques, and therapeutic ultrasound, 2 sessions per week for two weeks.
  Interventions: Other: myofascial induction and direct scar release techniques; Device: therapeutic ultrasound
- therapeutic ultrasound group (Experimental): They will receive a therapeutic ultrasound, 2 sessions per week for two weeks.
  Interventions: Device: therapeutic ultrasound

INTERVENTIONS:
Other: myofascial induction and direct scar release techniques — Manual therapy techniques used to reduce chronic lower transverse abdominal scars pain and improve quality of life of the affected women
  Arms: myofascial induction and direct scar release techniques group
Device: therapeutic ultrasound — Ultrasound petron (model SM 500) specifications: output frequency:1Mhz, output power:5W/cm², power intensity:5 degree (0.8-1.2-1.6-2.0-2.5), time intensity:5-30(step by 5 min) . It will be applied for both groups for 10 minutes

SUMMARY:
Postoperative scarring is one of the most common concerns among surgical patients. The incidence of abnormal scarring, i.e. keloid or hypertrophic scar formation after caesarean section (CS) is reported to be 41% .That can lead to functional limitations, pruritus, pain and cosmetic issues. so, the purpose of this study is to investigate quality of life and pain pressure threshold in response to myofascial induction and direct scar release techniques for lower transverse abdominal scar

DETAILED DESCRIPTION:
This study will be conducted on forty women with chronic lower transvers abdominal scar , they will be referred from department of Obstetrics and Gynecology ,Kasr Eleiny teaching Hospital and outpatient clinic of faculty of physical therapy, cairo university, Egypt.

All women will be randomly divided into two equal groups:

* Group A(Study group):It will include 20 women who will be treated by myofascial induction and direct scar release techniques in addition to therapeutic ultrasound, 2 sessions per week for two weeks.
* Group B(Control group):It will include 20 women who will be treated by therapeutic ultrasound, 2 sessions per week for two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women with a well healed, old , transverse cesarean section scar (more than 6 months resulted in chronic scar pain).
* Pain can be intermittent or constant at rest or with activity, and it is reported to be at least at a level of about 3/ 10 on visual analogue scale at recording sites will be marked on the C-section scar at 2.5 cm intervals (Wasserman et al., 2018).
* Women identified that the pain is either located in the cesarean section scar or caused by palpation of scar and it presents since the time of surgery not prior to the cesarean section.
* Their ages will range from 25-35 years old.
* Their BMI will be 18.5-29.9 kg/ m².

Exclusion Criteria:

* Acute and subacute cesarean section.
* Delayed wound healing.
* History of abdominal or pelvic cancer.
* Active pelvic or abdominal infection.
* Skin irritation/inflammation at the site of scar.
* Currently pregnant women.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-05 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Pain pressure threshold (PPT) | within 4 weeks
  * A pressure algometer will be used to measure pressure pain threshold for all participating women in both groups. ●
  * PPT recording sites will be marked on the C-section scar at 2.5 cm intervals. This resulted in from 5 to 8 measurement points along the scar.
  * Following, the marked points will be used to record PPTs in all time points for the PPT assessment; a 1-cm2 pressure probe will be positioned perpendicularly to the skin and pressed at a rate of 30kPa/s.Two measures will be collected for each area, with 30 seconds rest between point testing .
  * Average pressure pain threshold (pressure points across worst 3 points on scar averaged) will be used to analyze the PPT data .
scar mobility | within 4 weeks
  lower transverse abdominal scar mobility will be assessted by an adheremeter for both groups (A and B)before and after the end of treatment program.
  The adheremeter as described by Ferriero et al. has a radius of approximately 1.75 cm with concentric circles 2 mm apart . A mark will be made on the tightest part of the scar in four directions (superior, inferior, right and left). As there is no a contralateral side to abdominal tissue to be used as a reference range, we will use multi-directional scar mobility. Scar mobility measurements across the points will be averaged for each participating women and will be performed at the initial evaluation after 2 weeks (the end of the treatment) and at fourth week as follow up
Patient and Observer Scar Assessment Scale (POSAS) | within 4 weeks
  It includes subjective symptoms of pain and pruritus. It consists of 2 numerical numeric scales,it assesses vascularity, pigmentation, thickness, relief, pliability, and surface area, and it incorporates patient assessments of pain, itching, color, stiffness, thickness, and relief . The observer scar assessment scale rated five variables, each variable used a 10-point scoring system, summed to obtain a total score ranging from 5 to 50, with 5 representing normal skin with no associated symptoms. The patient scar assessment scale consisted of six items on scar-related pain, itchiness, color, stiffness, thickness, and irregularity. Each item used a 10-point scoring system, summed to obtain a total score ranging from 6 to 60, with 6 representing normal skin with no associated symptoms.

SECONDARY OUTCOMES:
quality of life assessment | within 4 weeks
  Short form 36 (SF-36) questionnaire will be used to assess the health-related quality of life .for all women in both groups (A and B)before and after the end of the treatment program.
  It measures health on eight multi-item dimensions, covering functional status, well-being, and overall health evaluation, each associated with 2-10 possible answers. The answer to each question is extrapolated to a standardized set of answers, and the results are transferred to a scale of 0-100, where 0 represents the worst state of health, and 100 represents the best state of health measured.

CONTACTS AND LOCATIONS:
Overall Officials: Manal M El-shafei, PHD, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF